CLINICAL TRIAL: NCT06561139
Title: Mindfulness as an add-on Intervention in Treatment for Problem Gambling - a Randomized Control Trial and a Qualitative Analysis in Clinical Settings in Sweden
Brief Title: Mindfulness as an add-on Intervention in Treatment for Problem Gambling in Clinical Settings in Sweden
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mindfulness gambling study
Record Dates: First submitted 2024-08-16; First posted 2024-08-19 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Problem Gambling
Keywords: Problem gambling; Mindfulness
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Randomized control trial, and subsequently a qualitative study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: treatment as usual + group mindfulness (Experimental): Eight-week, weekly group sessions of mindfulness, as an add-on to treatment as usual for problem gambling.
  Interventions: Behavioral: Mindfulness
- Control: treatment as usual + waiting list for two months (Active Comparator): Treatment as usual for problem gambling and waiting list for the mindfulness condition for two months, after which subjects are offered to undergo the same intervention as in the intervention group.
  Interventions: Behavioral: Mindfulness

INTERVENTIONS:
Behavioral: Mindfulness — Weekly group sessions of mindfulness, for eight weeks

SUMMARY:
This study will test the effects of an add-on mindfulness intervention for patients with gambling problems, added to treatment as usual, compared to a waitlist control condition. The study will primarily aim to decrease gambling behaviour compared to the control condition which receives the intervention later, after two months, and secondarily to decrease symptoms of depressive and anxiety symptoms. In addition, patients who have undergone the mindfulness intervention will be offered participation in a qualitative interview study aiming to deepen the understanding of feasibility and challenges of a mindfulness add-on intervention against gambling problems.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in any kind of treatment for problem gambling at a regional health care unit for problem gambling or at any municipal social service unit for problem gambling, and who provides informed consent

Exclusion Criteria:

* Inability to provide informed consent due to language difficulties or due to severe mental health problems, or because of mental health problems requiring urgent psychiatric management (such as suicidal, homicidal, delirious or psychotic behavior)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in past 30-day gambling (NODS 30 days) | Post-treatment (treatment completion) and 3 and 12 months after end of treatment
  Change in the number of criteria met according to a diagnostic tool for gambling disorder, but measuring the past 30 days at baseline and at post-treatment, and 3 and 12 months post-treatment

SECONDARY OUTCOMES:
Change in past-2-week depressive symptoms | Post-treatment (treatment completion) and 3 and 12 months after end of treatment
  Change in scores on Patient Health Questionnaire-9, a well-recognised instrument measuring past-2-week depressive symptoms
Change in past-2-week anxiety symptoms | Post-treatment (treatment completion) and 3 and 12 months after end of treatment
  Change in scores on Generalised Anxiety Disorder-7, a well-recognised instrument measuring past-2-week anxiety symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Malmö Addiction Center, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No